CLINICAL TRIAL: NCT06743386
Title: Pilot Study Evaluating the Combination of Endoscopic Ultrasound-Guided Radiofrequency and FOLFIRINOX in Locally Advanced Pancreatic Cancer
Brief Title: Pilot Study of EUS-Guided Radiofrequency and FOLFIRINOX in Advanced Pancreatic Cancer (RadioFAP )
Acronym: RadioFAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: French Society of Digestive Endoscopy (Other)
Responsible Party: Principal Investigator, Marc BARTHET, Director, Head of Endocopy, Principal Investigator, Medical doctor, French Society of Digestive Endoscopy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SFED-159
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: EUS-Guided Radiofrequency Ablation (RFA); Pancreatic Tumor Ablation; Minimally Invasive Tumor Treatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EUS-Guided Radiofrequency Ablation (RFA) (Experimental): Therapeutic procedure that combines endoscopic ultrasound (EUS) with radiofrequency ablation technology according to the practices of the investigating center
  Interventions: Device: Therapeutic procedure combines EUS-Guided Radiofrequency Ablation (RFA)

INTERVENTIONS:
Device: Therapeutic procedure combines EUS-Guided Radiofrequency Ablation (RFA) — It will be performed under general anesthesia with intubation, using a sectorial probe echoendoscope to target pancreatic tumors. Prophylactic measures, including intrarectal Diclofenac and antibiotics, are used to prevent complications. A high-frequency monopolar electrode needle is inserted into the lesion under ultrasound guidance, avoiding critical structures like pancreatic and biliary ducts. Energy is delivered until specific safety parameters are met, with multiple applications to maximize tumor coverage. RFA sessions are scheduled before, midway, and after chemotherapy cycles, and progress is monitored with routine imaging. Post-procedure care includes fasting, pain management, and standard blood tests. Patients are typically discharged the day after the procedure if no complications occur. Further treatment plans, including continuation or modification of chemotherapy and RFA, are determined based on disease progression observed in follow-up scans.

SUMMARY:
Pancreatic adenocarcinoma (PDAC) constitutes 90% of pancreatic tumors and is projected to become the second leading cause of cancer-related mortality in Europe by 2030. In France, its incidence doubled in men and tripled in women between 1982 and 2012. PDAC remains the digestive cancer with the poorest prognosis, with a five-year overall survival rate below 10% across all stages. Only surgical management with R0 resection (surgical margins free of cancer cells) offers a chance for cure or prolonged survival. However, surgery is feasible in only 15% of patients, as the disease is typically diagnosed at a late stage-locally advanced in 35% of cases or metastatic in 50%. Chemotherapy, specifically FOLFIRINOX, is the standard treatment for advanced cases, but resistance to chemotherapy poses a significant challenge. A key contributor to this resistance is the tumor stroma, which constitutes most of the tumor mass. This fibrous tissue acts as a mechanical barrier, restricting blood flow and potentially limiting the delivery of chemotherapy to cancer cells. The development of endoscopic ultrasound-guided radiofrequency ablation (EUS-RFA) has shown promise in treating pancreatic neuroendocrine tumors (pNETs) and pancreatic cystic neoplasms, sparking interest in its potential for PDAC. Preliminary studies demonstrate the feasibility of radiofrequency in PDAC, showing increased blood flow around treated sites. Combining systemic chemotherapy with radiofrequency may enhance drug diffusion and improve treatment efficacy. Additionally, tumor thermoablation could stimulate an immune response, as observed in experimental and clinical research. This study aims to evaluate the feasibility of tumor destruction via radiofrequency ablation combined with FOLFIRINOX in improving progression-free survival for patients with PDAC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 18
2. Patients with locally advanced, borderline resectable, or inoperable pancreatic adenocarcinoma, confirmed by histological or cytological tests and assessed through a multidisciplinary consultation.
3. Patients without evidence of metastases.
4. No prior anti-tumoral treatment.
5. World Health Organization (WHO) performance status ≤ 1.
6. Measurable tumor according to the RECIST v1.1 criteria: a tumor lesion with the largest diameter ≥ 20 mm using conventional imaging techniques or ≥ 10 mm using spiral CT scan.
7. Patient who has provided written consent.
8. Patient with no contraindications to general anesthesia.
9. Pancreatic tumor accessible via endoscopic ultrasound.
10. Patient enrolled in a social security program (beneficiary or dependent).

Exclusion Criteria:

* 1. Other types of non-ductal or solid pancreatic tumors, including endocrine tumors, acinar cell adenocarcinoma, cystadenocarcinoma, and malignant ampullary tumors.

  2. Presence of metastases. 3. Contraindication to treatment with 5FU, oxaliplatin, or irinotecan. 4. Patients with a tumor that could benefit from neoadjuvant treatment with radiochemotherapy or chemotherapy alone for secondary resection (decision by a multidisciplinary committee).

  5. Pre-existing neuropathy, Gilbert's disease, or known UGT1A1*28/*28 genotype. 6. Chronic inflammatory bowel disease. 7. Other concurrent cancers, or a history of cancer within the last 5 years, except for in situ cervical cancer that has been treated or a properly treated basal cell carcinoma or squamous cell carcinoma.

  8. Hereditary intolerance to fructose. 9. Individuals deprived of liberty or under guardianship. 10. Inability to follow up with the study due to geographical, social, or psychological reasons.

  11. Contraindication to echo-endoscopy-guided cytopuncture (coagulation disorders or previously operated stomach).

  12. Neutrophil count < 1500/mm³. 13. Platelet count < 70,000/mm³. 14. Patients are not effectively treated for neoplastic jaundice if present at diagnosis.

  15. Patient in an exclusion period or currently participating in another clinical research protocol.

  16. Patients are unable to understand or read the information/consent form. 17. Pregnant women or those wishing to become pregnant during the study period, or breastfeeding women.

  18. Patients with implanted pacemakers or implantable cardioverter-defibrillators (ICDs).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
The success rate of tumor destruction achieved using radiofrequency ablation (RFA) with a radiofrequency needle guided by endoscopic ultrasound (EUS), in combination with chemotherapy. | 2, 6, 9, 12, and18 months
  This rate will be defined as the ratio of satisfactory deliveries (without serious adverse events) to the total number of deliveries performed

SECONDARY OUTCOMES:
Progression-Free Survival: | 2, 6, 9, 12, and18 months
  The time interval between the date of enrollment in the study and the point at which the disease progresses
Impact of radiofrequency tumor ablation combined with FOLFIRINOX on overall survival | 2, 6, 9, 12, and18 months
  Measured from study enrollment to date of death, regardless of cause
Impact of radiofrequency tumor ablation with FOLFIRINOX on quality of life | 2, 6, 9, 12, and 18 months
  Assessed using the EORTC QLQ-C30 questionnaire
Effect of radiofrequency ablation combined with FOLFIRINOX on secondary resectability | 2, 6, 9, 12, and18 months
  Assessed through regular CT scans (RECIST 1.1) to determine if initially unresectable tumors become resectable after RFA treatment
Pancreatic intratumoral radiofrequency technical success | 14 days before chemotherapy and at 2 and 4 months post-treatment.
  Defined as successful EUS-RFA execution, including needle insertion and ablation feasibility
RFA tolerance | 14 days before chemotherapy and at 2 and 4 months post-treatment.
  Defined as the ratio of adverse events (AEs) to the total number of patients who underwent EUS-RFA